CLINICAL TRIAL: NCT06855108
Title: Caffeine for Hypoxic Ischemic Encephalopathy (CHIME Trial)
Brief Title: Caffeine for Hypoxic Ischemic Encephalopathy
Acronym: CHIME
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: RTI International (Other); University of North Carolina, Chapel Hill (Other); Kinshasa School of Public Health (Other); Institute of Nutrition of Central America and Panama (INCAP) (Unknown); Lata Medical Research Foundation, Nagpur (Other); Aga Khan University (Other); University Teaching Hospital, Lusaka, Zambia (Other); KLE Academy of Higher Education and Research (Deemed- to- be-University), Jawaharlal Nehru Medical College (JNMC), Belagavi, India (Unknown); Bill and Melinda Gates Foundation (Other); University of Virginia (Other); University of Alabama at Birmingham (Other); Thomas Jefferson University (Other); Columbia University (Other); University of Colorado, Denver (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP CHIME; INV-068776 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2025-01-27; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hypoxic Ischemic Encephalopathy (HIE)
Keywords: Caffeine; Hypoxic Ischemic Encephalopathy; HIE; AKI
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: 1:1 individually randomized, parallel-arm, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The protocol study team, international principal investigator (iPI), site staff and participants will be masked to the assigned treatment arm. Lab personnel will be masked to the assigned treatment arm until assays for samples collected after randomization are complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine citrate oral solution (Experimental): Participants randomized to the oral caffeine arm will receive a single 20 mg/kg loading dose of caffeine citrate administered enterally within 6 hours after delivery, followed by a 10 mg/kg dose every 24 hours for two additional doses.
  Interventions: Drug: Caffeine citrate oral solution
- Oral placebo (Placebo Comparator): Participants randomized to the oral placebo arm will receive a single identical placebo administered enterally within 6 hours after delivery, followed by an identical placebo dose every 24 hours for two additional doses.
  Interventions: Drug: Oral placebo solution

INTERVENTIONS:
Drug: Caffeine citrate oral solution — Caffeine citrate oral solution will be used and administered by enteral route (oral or by gavage tube). The loading dose (20 mg/kg) will be administered once followed by daily doses of 10 mg per kg body weight every 24 hours for two doses. The study Standard Operating Procedures (SOPs) includes details regarding caffeine preparation based on the participant's body weight.
  Arms: Caffeine citrate oral solution
Drug: Oral placebo solution — Identical placebo oral solution
  Other Names: Oral placebo
  Arms: Oral placebo

SUMMARY:
CHIME is a randomized, parallel-arm, double-blind, placebo-controlled trial focused on infants with hypoxic ischemic encephalopathy (HIE). The trial will recruit neonates who are diagnosed with HIE within six hours after birth based on physiologic criteria (acidosis noted on an umbilical cord or early [<1 hour] postnatal blood sample) and neurologic criteria (modified Sarnat exam consistent with encephalopathy). Following informed consent, and by six hours after birth, neonates with HIE will be randomized to one of two treatment arms and subsequently receive one 20 mg/kg dose of oral caffeine followed by two additional 10 mg/kg doses at 24-hour intervals or placebo of the same regimen (three total doses).

The goal of this clinical trial is to compare the incidence of all-cause mortality OR moderate to severe neurodevelopmental impairment (NDI) at 18-22 months between neonates with HIE who are randomized to oral caffeine or placebo. Our hypothesis is that neonates with HIE who receive oral caffeine will have 10% lower incidence of all-cause mortality or moderate to severe NDI at 18-22 months compared to placebo.

DETAILED DESCRIPTION:
Background: One million newborns die annually due to intrapartum-related events (formerly referred to as birth asphyxia). Among survivors, intrapartum related events often lead to organ dysfunction with lasting consequences, including severe morbidity and neurodevelopmental impairment (NDI). Newborns exposed to significant intrapartum-related events can have brain injury, referred to as hypoxic ischemic encephalopathy (HIE). HIE is routinely treated with therapeutic hypothermia. However, a recent multi-national randomized controlled trial demonstrated that therapeutic hypothermia increased mortality from HIE in some contexts. Therefore, there is an urgent, unmet public health need to develop effective strategies for the treatment of HIE to prevent morbidity and mortality. Caffeine, a low-cost, readily available medication is a promising strategy for treatment of HIE given its neuroprotective, anti-inflammatory, and anti-oxidative properties. Furthermore, caffeine might have physiologic benefits beyond HIE, because a single dose of a methylxanthine (caffeine's drug class) reduces acute kidney injury in infants with HIE in settings where therapeutic hypothermia is not available.

Objective: To compare the incidence of all-cause mortality OR moderate to severe NDI at 18-22 months between neonates with HIE who are randomized to oral caffeine or placebo.

Hypothesis: Neonates with HIE who receive oral caffeine will have 10% lower incidence of all-cause mortality or moderate to severe NDI at 18-22 months compared to placebo.

Study Design: 1:1 individually randomized, parallel-arm, double-blind, placebo-controlled trial

Population: ≥ 36 week gestation and ≥1800 grams liveborn neonates who meet both physiologic and neurologic criteria for moderate to severe HIE and live in the Global Network research sites

Intervention: The intervention arm will receive one 20 mg/kg loading dose of caffeine given within 6 hours of delivery, followed by a daily dose of 10 mg/kg, given every 24 hours for 2 doses (total of 3 doses).

Comparison: The comparison arm will receive placebo using an identical dosing regimen.

Primary outcomes: All-cause mortality or moderate to severe NDI at 18-22 months of age

Sub-Studies: In conjunction with the CHIME Trial, we will embed 3 sub-studies to be conducted within subsets of CHIME participants. A sample will be chosen by convenience for each sub-study.

Pharmacokinetics Sub-study: For approximately 40 participants per Global Network research site, we will collect 2-3 blood samples during the birth hospitalization for pharmacokinetic (PK) analysis of caffeine. We will use a population PK approach to characterize the PK of infants with HIE, and to relate caffeine exposure to mortality or moderate to severe disability.

Neuro-imaging Sub-Study: For participants who are born at or follow-up in a facility with the capability of performing ultra-low-field (ULF) magnetic resonance imaging (MRI), we will obtain ULF MRI brain images during the birth hospitalization and at the 6-month follow-up visit. We will relate the findings on ULF MRI to the severity of HIE at enrollment and to the neurodevelopmental outcomes.

Omics Sub-Study: For participants for whom cord blood is available, we will obtain a sample of cord blood to be stored for future multi-omic analyses (e.g., genomic, transcriptomic, proteomic, and metabolomic). We will use multi-omics to identify molecular signatures associated with HIE.

ELIGIBILITY:
Participant Inclusion Criteria:

Infants who meet all the following criteria are eligible for enrollment as study participants:

1. Liveborn infants ≥36 weeks
2. Birth weight ≥1800 grams
3. Meets physiologic criteria for moderate to severe HIE, defined as meeting either of the following two criteria:

   1. Criterion #1: Severe acidosis, defined as an umbilical cord sample or neonatal serum sample within one hour after birth demonstrating any of following criteria:

      * pH <7.0; or
      * Base Deficit ≥16 mmol/L; or
      * Lactate >8 mmol/L.
   2. Criterion #2: Participant must meet all of the following three criteria:

   i. Moderate acidosis, defined as an umbilical cord sample or neonatal serum sample within one hour after birth demonstrating any of following criteria:
   * POC pH 7.0-7.15; or
   * Base Deficit 10.0-15.9 mmol/L; or
   * Lactate 6-8 mmol/L.

   ii. Evidence of an acute perinatal event (i.e., placental abruption, intrapartum hemorrhage, cord prolapse, severe fetal heart rate abnormality, uterine rupture).

   iii. Any of the following criteria:
   * 10-minute Apgar <5; or
   * Need for assisted ventilation initiated at birth and continued for ≥10 minutes
4. Meets neurologic criteria for moderate to severe HIE, defined as a physical exam conducted between one and six hours after birth that meets either of the following criteria:

   1. Moderate to severe encephalopathy in at least three out of six modified Sarnat categories (level of consciousness, spontaneous activity, muscle tone, posture, primitive reflexes, autonomic function); or
   2. A clinical diagnosis of seizure in the first six hours after birth.

Participant Exclusion Criteria:

Infants who meet any of the following criteria are not eligible for enrollment as study participants:

1. Home births
2. Infants who cannot be enrolled, randomized and receive study medication within 6 hours post-delivery
3. Infants with a recognized major congenital anomaly or genetic syndrome that would affect their neurodevelopment.
4. Infants for whom medical care will not be provided based on the severity of their condition or any other condition that would preclude participation per clinical judgement.
5. Infant has received therapeutic hypothermia or there is a clinical plan to initiate active or passive hypothermia for the infant.
6. Infants who will be unavailable to complete follow-up visits.
7. Infants who have received caffeine after delivery.
8. Infants whom the health care team deem ineligible for the study based on likelihood to receive caffeine outside of the study protocol.
9. Enrollment in another trial that will impact participation in this trial.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 830 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Composite outcome, defined by the occurrence of any of the following: | 18-22 months
  All-cause infant mortality or moderate to severe neurodevelopmental impairment

SECONDARY OUTCOMES:
Secondary composite outcome, defined by the occurrence of any of the following: | 18-22 months
  All-cause infant mortality or severe neurodevelopmental impairment
All-cause neonatal mortality | 28 days after delivery
  Death from any cause to 28 days after delivery
All-cause infant mortality | 12 months
  Death from any cause before first birthday
All-cause mortality | 18 months
  Death from any cause
Time to all-cause mortality | 18-22 months
  Timespan from randomization to death from any cause
Severe neurodevelopmental impairment | 18-22 months
Moderate neurodevelopmental impairment | 18-22 months
Composite cognitive, language, and motor scores on the Bayley Scales of Infant and Toddler Development-Fourth Edition | 18-22 months
  Cognitive Scale on the Bayley Scales of Infant and Toddler Development - Fourth Edition
  - Scale ranges from 55-145 such that higher scores indicate a better cognitive outcome.
  Language Scale on the Bayley Scales of Infant and Toddler Development - Fourth Edition - Scale ranges from 45-155 such that higher scores indicate a better language outcome.
  Motor Scale on the Bayley Scales of Infant and Toddler Development - Fourth Edition
  - Scale ranges from 45-155 such that higher scores indicate a better motor outcome.
Hammersmith Infant Neurological Exam score | 6 months
  Ranges from 0 to 78 where higher scores indicate a better neurological outcome.
Global Scale for Early Development D-score and DAZ | 12 months
  Global Scale for Early Development D-score: Ranges from 0 to 100 where higher scores indicate a higher level of overall development.
  Global Scale for Early Development DAZ: Ranges from -5 to 5 where higher scores indicate a higher level of overall development.
Global Scale for Early Development Short Form D-score and DAZ | 18-22 months
  Global Scale for Early Development D-score: Ranges from 0 to 100 where higher scores indicate a higher level of overall development.
  Global Scale for Early Development DAZ: Ranges from -5 to 5 where higher scores indicate a higher level of overall development.
Acute kidney injury within the first postnatal week | Postnatal days 2-4
  Defined as an increase in serum creatinine of 0.3 mg/dL or more on 2 measurements
Manual blood pressure (systolic and diastolic) | 18-22 months
  Systolic and diastolic blood pressure taken using manual measurement
Hypertension | 18-22 months
  Based on the systolic blood pressure at the ≥95% for age related normative values
Serum creatinine | 18-22 months
  Measured using serum creatinine testing.
Serious adverse events (SAEs) | Discharge or 7 days after administration of the last study drug (whichever occurs first)
  An SAE form will be completed for any event meeting the following criteria:
  * Results in participant death;
  * Is life-threatening;
  * Requires hospitalization or prolongs existing hospitalization;
  * Results in persistent or significant disability or incapacity;
  * Any other serious or unexpected AE that the study investigator(s) feels should be reported.
Adverse events of special interest (AESIs) | Discharge or 7 days after administration of the last study drug (whichever occurs first)
  To include:
  * Clinically diagnosed seizures
  * Receipt of any antiepileptic drug
  * Seizures not controlled on one antiepileptic drug
  * Hypoglycemia (BG <30 mg/dL)
  * Hyperglycemia (BG >200 mg/dL)
  * Heart rate [HR] >180 beats per minute [bpm] within 30 minutes of study drug administration
  * Necrotizing enterocolitis (NEC): as defined by feeding intolerance, bloody stool and abdominal distension
Length/height and length/height-for-age z-score | Birth, 1 month, 6 months, 12 months, and 18-22 months
  Length/height and length/height-for-age z-score
Weight and weight-for-age z-score | Birth, 1 month, 6 months, 12 months, and 18-22 months
  Weight and weight-for-age z-score
Head circumference and Head circumference-for-age z-score | Birth, 1 month, 6 months, 12 months, and 18-22 months
  Head circumference and Head circumference-for-age z-score

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Bauserman, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Elizabeth M McClure, PhD, Principal Investigator — RTI International; Denise C Babineau, PhD, Principal Investigator — RTI International
Locations (7):
- ICDDR,B, Saidpur, Bangladesh
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Institute of Nutrition of Central America And Panama (INCAP), Chimaltenango, Guatemala
- India (2):
  - KLE University's J N Medical College, Belagavi
  - Lata Medical Research Foundation, Nagpur
- Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
Only aggregate and deidentified data will be shared.